CLINICAL TRIAL: NCT00393822
Title: A Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Palifermin (Recombinant Human Keratinocyte Growth Factor) for Reduction of Oral Mucositis in Subjects With Stage 2B or 3 Locally Advanced, Colon Cancer Receiving 5-FU and Leucovorin as Adjuvant Therapy
Brief Title: A Study of Palifermin for the Reduction of Oral Mucositis in Subjects With Stage 2B or 3 Locally Advanced, Colon Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 20040122
Record Dates: First submitted 2006-10-26; First posted 2006-10-30 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Colon Cancer
Keywords: KGF; Palifermin; Oral Mucositis; Clinical Trial; Amgen; Oncology; Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms; Stomatitis; Neoplasms | interventions — Fibroblast Growth Factor 7

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palifermin (Experimental): 50 subjects to receive palifermin 3 days prior to the first day (day 1) of each cycle of 5-FU/ LV chemotherapy.
  Interventions: Drug: palifermin
- Control Group (Placebo Comparator): 50 subjects to receive matched placebo 3 days prior to the first day (day 1) of each cycle of 5-FU/ LV chemotherapy.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: palifermin — dose of 120 μg/kg, intravenous (IV) on day -3 for each cycle, for up to 6 chemotherapy cycles
  Other Names: KGF
  Arms: Palifermin
Drug: placebo — one bolus IV injection at 120 μg/kg/day of matched placebo
  Other Names: Pbo
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of palifermin (recombinant human keratinocyte growth factor, rHuKGF) in reducing the incidence of oral mucositis in subjects with stage 2B and 3 locally advanced, colon cancer receiving chemotherapy as an adjuvant treatment for their disease.

DETAILED DESCRIPTION:
This study is being conducted to determine whether administration of a single IV dose of palifermin 3 days before initiation of chemotherapy and 3 days before each subsequent treatment cycle would reduce the incidence of oral mucositis and to evaluate the safety profile in the subject population. This study will evaluate the efficacy of palifermin in reducing the incidence of grade ≥ 2 OM in subjects with stage 2B or stage 3 locally advanced, colon cancer undergoing adjuvant chemotherapy with 5-FU and leucovorin in cycle 1. This study will also assess the safety and tolerability of palifermin administered as a single IV dose before each cycle of 5-FU and leucovorin, evaluate the effect of palifermin on patient-reported mouth and throat soreness, the incidence of grade ≥ 2 oral mucositis in cycle 2, the duration of grade ≥ 2 oral mucositis, 5-FU dose reductions/delays and the long-term effects of palifermin on disease outcome and survival.

ELIGIBILITY:
Inclusion Criteria:

* History of newly diagnosed histologically confirmed resected colon cancer (American Joint Committee on Cancer [AJCC] Stage 2B or 3) and a candidate for adjuvant 5-FU and Leucovorin
* Eastern Cooperative Oncology Group performance status ≤ 1
* Functional hematopoietic and hepato-renal systems

Exclusion Criteria:

* Previous therapy (e.g. chemotherapy, radiotherapy or biological therapy) for colon cancer, other than surgical tumor resection
* Presence or history of any other primary malignancy
* Presence of active or chronic oral mucositis or xerostomia
* Previous treatment with other keratinocyte growth factors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-08; Primary Completion 2007-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Grade ≥ 2 (WHO scale) oral mucositis | in Cycle 1 of chemotherapy treatment phase

SECONDARY OUTCOMES:
Incidence of chemotherapy (5-FU) dose reductions and dose delays | in Cycle 2 of chemotherapy treatment phase
Average mouth and throat soreness (MTS) score | in Cycle 1 and in Cycle 2 of chemotherapy treatment phase
Duration of grade ≥ 2 (WHO scale) oral mucositis | in Cycle 1 and in Cycle 2 of chemotherapy treatment phase
Incidence and severity of adverse events | during Treatment Phase (6 cycles of chemotherapy)
Changes in laboratory values | during Treatment Phase (6 cycles of chemotherapy)
Incidence of serum anti-palifermin antibody formation | during Treatment Phase (6 cycles of chemotherapy)
Progressive disease rate | at 6 months
Incidence of secondary primary tumors | within long-term follow-up phase
Incidence of other malignancies | within long-term follow-up phase
Progression-free survival (PFS) | within long-term follow-up phase
Overall survival (OS) | within long-term follow-up phase
Incidence of grade ≥ 2 (WHO scale) oral mucositis | in Cycle 2 of chemotherapy treatment phase

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_24_KGF_20040122.pdf
- See also: FDA-approved Drug Labeling — http://www.kepivance.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com